CLINICAL TRIAL: NCT06413043
Title: Study on Efficacy of Add on Selenium in Mild-to-moderate Graves Ophthalmopathy: A Randomized Control Trial
Brief Title: Study on Efficacy of Add on Selenium in Mild-to-moderate Graves Ophthalmopathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, Sandip Kumar Sahu, Associate Professor, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PG Thesis/2023-24/122
Record Dates: First submitted 2024-04-29; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Thyroid Eye Disease; Graves Ophthalmopathy
Keywords: Thyroid Eye Disease; Graves Ophthalmopathy
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — Selenium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADD on Selenium (Active Comparator): Add on Selenium (100mcg once daily) with Vitamin B Complex and Standard Treatment for Grave's Disease
  Interventions: Drug: Selenium
- Placebo (No Intervention): Vitamin B Complex supplementation with Standard Treatment for Grave's Disease

INTERVENTIONS:
Drug: Selenium — Add on Selenium (100mcg once daily) with Vitamin B Complex and Standard Treatment for Grave's Disease
  Arms: ADD on Selenium

SUMMARY:
The Study on efficacy of add on selenium in mild-to-moderate Graves ophthalmopathy: A Randomized Control Trial.; The study aims to evaluate the response of adding selenium in patients with Graves ophthalmopathy, focusing on improving quality of life, CAS scoring, and thyroid status. The methodology involves a Randomized Control Trial with a sample size of 78 patients. Patients meeting specific criteria will receive either standard treatment with Anti Thyroid Drugs and Vitamin B complex or add on selenium with Vitamin B complex for 6 months. Outcome measures include CAS score reduction, thyroid function improvement, and quality of life enhancement. The study will last 18 months, with various investigations and ethical considerations outlined. The document emphasizes the importance of early diagnosis of Graves Ophthalmopathy to prevent vision loss and deformity, highlighting the significance of informed patients and healthcare professionals regarding TED symptoms and risk factors.

DETAILED DESCRIPTION:
The Study on efficacy of add on selenium in mild-to-moderate Graves ophthalmopathy: A Randomized Control Trial. The study aims to evaluate the response of adding selenium in patients with Graves ophthalmopathy, focusing on improving quality of life, CAS scoring, and thyroid status. The methodology involves a Randomized Control Trial with a sample size of 78 patients. Patients meeting specific criteria will receive either standard treatment with Anti Thyroid Drugs and Vitamin B complex or add on selenium with Vitamin B complex for 6 months. Outcome measures include CAS score reduction, thyroid function improvement, and quality of life enhancement. The study will last 18 months, with various investigations and ethical considerations outlined. The document emphasizes the importance of early diagnosis of Graves Ophthalmopathy to prevent vision loss and deformity, highlighting the significance of informed patients and healthcare professionals regarding TED symptoms and risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Mild-to-moderate Grave's Ophthalmopathy in Age group >18years

With only one or more :

* Retraction of lid <2 mm
* Mild soft tissue involvement
* Proptosis of <=3 mm
* Corneal exposure that responds to lubricating eyedrops.
* Patients with CAS < = 4
* Patients diagnosed with hyperthyroidism converted to euthyroid since 2 months with Anti Thyroid Drugs.
* Those who are willing to follow the advised treatment and timely follow ups.

Exclusion Criteria:

* Treatment with any steroid (Intravenous, oral or topical) for any condition within 3 weeks before presentation.
* Any treatment with rituximab
* Any earlier treatment with teprotumumab.
* Any treatment with monoclonal antibody within 3months before presentation.
* Lactating or pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-05-06 (Estimated); Primary Completion 2025-08-05 (Estimated); Study Completion 2025-11-05 (Estimated)

PRIMARY OUTCOMES:
To evaluate and compare the response of add on selenium in patients with grave's ophthalmopathy | 90 Days
  To evaluate and compare the response of add on selenium in patients with grave's ophthalmopathy, with Best corrected visual Acuity, Clinical activity Score (CAS ), Increase in measured proptosis (bulging of the eyes) > 2 mm over 1-3 months. Decrease in eye movement limit of > 8° over 1-3 months. Decrease in visual acuity (2 Snellen chart lines) over 1-3 months. A CAS score greater than 4 is associated with active disease. The positive predictive value of CAS > 4 is approximately 80%, and the negative predictive value is around 64%

SECONDARY OUTCOMES:
the effects of Grave's ophthalmopathy on Patient's perception of their position in life in the context of the culture and value systems in which they live and in relation to their goals, expectations, standards and concerns | 90 Days
  To study the effects of Grave's ophthalmopathy on Patient's perception of their position in life in the context of the culture and value systems in which they live and in relation to their goals, expectations, standards and concerns, through the World Health Organization Quality of Life Brief Version- Brief(WHOQOL-BRIEF) questionnaire.
  The 4 domain scores are each converted into a scale from 0 to 100. For this purpose, the number 4 is subtracted from each of the domain scores, and the difference is multiplied by 100/16 or the number 6.25. 0 points represent the worst possible state of health, while 100 points represent the best possible state of health with regard to the respective domain. Thus, the patient's physical, psychological, social, and environmental state of health are assessed separately.
To Assess the Colour Vison | 90 Days
  Anomaloscopes are optical instruments in which the observer must manipulate stimulus control knobs to match two colored fields in color and brightness.
  Measurement Unit: Typically, color vision is assessed qualitatively (normal or deficient).
  Minimum Value: Normal color vision (able to perceive a wide range of colors). Maximum Value: Color vision deficiency (varies based on the type of deficiency).
To Assess the Fundus | 90 Days
  Fundus Examination:
  Measurement Unit: No specific unit; it's a visual assessment. Minimum Value: Normal fundus appearance (no abnormalities). Maximum Value: Various abnormalities (e.g., diabetic retinopathy, hypertensive retinopathy).
To Examine Thyroid Function Test | 90 Days
  Thyroid Function Test:
  TSH: Normal range is approximately 0.4 to 4.0 μIU/mL. T4: Normal range is around 4.5 to 11.2 μg/dL. T3: Normal range varies but is generally 80 to 200 ng/dL

CONTACTS AND LOCATIONS:
Locations (1):
- AIIMS Bhubaneswar, Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bartalena L, Tanda ML. Current concepts regarding Graves' orbitopathy. J Intern Med. 2022 Nov;292(5):692-716. doi: 10.1111/joim.13524. Epub 2022 Jun 1. PMID 35604323
- [Result] Burch HB, Perros P, Bednarczuk T, Cooper DS, Dolman PJ, Leung AM, Mombaerts I, Salvi M, Stan MN. Management of thyroid eye disease: a Consensus Statement by the American Thyroid Association and the European Thyroid Association. Eur Thyroid J. 2022 Dec 8;11(6):e220189. doi: 10.1530/ETJ-22-0189. Print 2022 Dec 1. PMID 36479875
- [Result] Lanzolla G, Marino M, Marcocci C. Selenium in the Treatment of Graves' Hyperthyroidism and Eye Disease. Front Endocrinol (Lausanne). 2021 Jan 26;11:608428. doi: 10.3389/fendo.2020.608428. eCollection 2020. PMID 33574798